CLINICAL TRIAL: NCT05985447
Title: Menopause Related Influences on Leukocyte Distribution, Monocyte Function and Platelet Reactivity
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: Hormone
Record Dates: First submitted 2023-04-14; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Arteriosclerosis; Acute Myocardial Infarction; Cardiovascular Events; Menopause
Keywords: sex; gender; female; male; menopause; hormone replacement therapy; Atherosclerosis; cardiovascular events; cardiovascular risk
MeSH Terms: conditions — Arteriosclerosis; Coitus; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — prospectively defined blood sampling protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Women and men show marked differences in cardiovascular risk profile and outcome. Women experience fewer cardiovascular events than men before menopause, but this relationship seems to reverse at menopause. These disparities are probably due to hormonal factors, especially the female sex hormone estrogen seems to have a protective influence on the development of atherosclerotic plaques premenopausal.

The underlying mechanisms of the effect of estrogens on the vessel wall are still insufficiently investigated. In this study, menopause related effects on leukocyte distribution and function as well on platelets and their aggregational response will be evaluated.

DETAILED DESCRIPTION:
Sex-specific differences in the risk profile and outcome of cardiovascular diseases are evident, which are probably due to hormonal factors. Women suffer significantly fewer cardiovascular events than men before menopause, after menopause this relationship seems to reverse. Moreover, outcome is worse in female patients compared to men.

Platelets and leukocytes play an essential role in cardiovascular risk. Nevertheless, the underlying mechanisms of the mechanistic effects of the hormone transition in menopause on leukocytes and platelets have only been insufficiently investigated so far. Moreover, effects of a possible hormone replacement therapy are insufficiently understood with contradictive literature concerning cardiovascular effects.

The aim in this study, is to analyse leukocyte and platelet function in dependence from menopause related changes in hormone levels of estrogen, testosterone, progesterone, LH and FSH. Moreover, hormone replacement therapy will be investigated.

For this purpose, blood samples from male and female patients will be investigated with regard to age and menopause status. The blood samples are analysed by FACS to differentiate the leukocytes and test for inflammatory properties and reactive oxygen species. The monocyte distribution divided according to the surface markers CD14 and CD16 is analysed. In addition, plasma from the patient samples will be used to assess hormone levels in the blood. In addition, patient data such as general laboratory parameters, risk and lifestyle factors are collected and associated with the hormone and lipid levels.

For platelet function analysis, light-transmittance aggregometry, flow cytometry (platelet leukocyte crosstalk, investigation of platelet surface markers for platelet activation and cell-cell-adhesion) will be investigated. Platelets secretory potency will be analysed by ATP-release. Moreover, platelet adhesion will be investigated by collagen-coated flow chambers. Platelet proteomics and RNA sequencing will complement the data in an unbiased approach. In addition in-vitro incubation analyses with estrogen and testosterone will be conducted to investigate hormone replacement therapy effects.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Male, female, diverse patients with current treatment in the Department of Cardiology, Pneumology and Angiology.
* Persons who are able to understand and follow the instructions of the study staff
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Lack of written consent to participate in the study
* coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female Patients with and without cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Leukocyte distribution measured by flow cytometry | single time, up to one day after inclusion
  CD45 (Leukocytes), CD3 (T-cells), CD14 (Monocytes), CD16 (Granulocytes), CD19 (B-cells)
Platelet function | single time, up to one day after inclusion
  measured by light transmittance aggregometry (Parameters: Maximum of Aggregation, Slope
Platelet surface markers, platelet leukocyte crosstalk (CD40, CD40L) | single time, up to one day after inclusion
  measured by flow cytometry (FACS)

SECONDARY OUTCOMES:
Reactive Oxygen Species (ROS) Generation via CellRoxGreen [geometric mean] | single time, up to one day after inclusion
  measured by Flow Cytometry (FACS)
Hormone levels of estrogen | single time, up to one day after inclusion
  measured by ELISA [ng/l]
Hormone levels of testosterone measured by ELISA | single time, up to one day after inclusion
  measured by ELISA [ng/l]
Hormone levels of progesterone | single time, up to one day after inclusion
  measured by ELISA [µg/l]
Hormone levels of follicle stimulating hormone | single time, up to one day after inclusion
  measured by ELISA [µg/l]
Hormone levels of luteinizing hormone | single time, up to one day after inclusion
  measured by ELISA [µg/l]
Questionnaire including lifestyle factors, cardiovascular risk factors | single time, up to one day after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf
Locations (1):
- University-Hospital Düsseldorf Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No